CLINICAL TRIAL: NCT02105051
Title: A Population-based Investigation of Related Factors of Birth Weight in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Neonatal Network (Other)
Responsible Party: Principal Investigator, Chao Chen, director of neonatal department in Children's hospital of Fudan University ,professor,Chairman of Chinese neonatal network, Chinese Neonatal Network
Other Study IDs: ChNN-001
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Risk Factors; Birth Weight
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish Chinese neonatal network to investigate current situation of neonatal birth weight and related factors. We investigated the risk factors such as sex, gestational age, region, nation, altitude, place of residence, maternal occupation, education level of mother, maternal age, maternal pregnancy diseases and multiple births.

ELIGIBILITY:
Inclusion Criteria:

* live births
* Gestational age between 24 weeks and 43 weeks

Exclusion Criteria:

* Major malformation
* Physical deformity
* Fetal edema
* Body mass diagnosed in prenatal ultrasound
* Acute blood loss during delivery

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We continuously collected the information of live births in participating hospitals of Chinese neonatal network during the study period
Sampling Method: Non-Probability Sample
Dates: Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
birth weight | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan University, Shanghai, China